CLINICAL TRIAL: NCT06010329
Title: A Multicenter, Open-label, Phase 2 Study to Evaluate the Efficacy and Safety of Sutetinib Maleate Capsule in Locally Advanced or Metastatic NSCLC (Uncommon EGFR Mutations Only)
Brief Title: A Study to Evaluate the Efficacy and Safety of Sutetinib Maleate Capsule in Locally Advanced or Metastatic NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Teligene US (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TL-EGFR-2201
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Oncology; Sutetinib Maleate Capsule; Teligene; Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm, Open label (Experimental): Participants will receive sutetinib maleate capsule taken orally with (preferred) or without food, at the dose directed by the Investigators, 28 days for a cycle.
  Interventions: Drug: Sutetinib Maleate Capsule

INTERVENTIONS:
Drug: Sutetinib Maleate Capsule — Oral administration

SUMMARY:
The main objective of the study will be to evaluate the efficacy of sutetinib maleate capsules in participants with locally advanced or metastatic non-small cell lung cancer NSCLC (uncommon EGFR mutations only).

DETAILED DESCRIPTION:
Sutetinib is an investigational irreversible EGFR tyrosine kinase inhibitor. EGFR is a gene that makes a protein that is involved in cell growth and cell survival. Mutated (changed) forms of the EGFR gene and protein have been found in some types of cancer, including non-small cell lung cancer. These changes may cause cancer cells to grow and spread in the body. The purpose of this study is to explore how effective sutetinib maleate capsules are for the treatment of patients with locally advanced or metastatic NSCLC with uncommon EGFR mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old and above, male or female
2. Histopathological and/or cytopathological confirmation of locally advanced or metastatic NSCLC
3. Confirmation that the tumor harbors an uncommon epidermal growth factor receptor (EGFR) mutation (tumor tissue biopsy)
4. At least one measurable lesion
5. Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2
6. A minimum life expectancy of > 3 months
7. Adequate bone marrow reserve, hepatic, renal, and coagulation function

Other inclusion criteria apply for participating in the study.

Exclusion Criteria:

1. Participant ever used the epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR TKI) for anti-tumor therapy prior to enrollment (Cohort 1), or second generation EGFR TKI (Cohort 2)
2. Any systemic anti-tumor therapy such as chemotherapy and radiation therapy (including curative radiotherapy or spinal radiotherapy portion >30%) used within 3 weeks prior to enrollment; immunotherapy within 4 weeks; any palliative radiotherapy for non-target lesions used to relieve symptoms and traditional Chinese medicines indicated for the tumor within 2 weeks prior to enrollment; Cohort 2: any EGFR TKIs within 5 half-lives.
3. Use or intake of drugs or foods containing potent inhibitors or inducers of cytochrome P450 isozyme 3A4 (CYP3A4) within 14 days or 5 half-lives, whichever is the longer, prior to enrollment
4. Surgical operation (excluding aspiration biopsy) of main organs or a significant injury within 4 weeks prior to enrollment
5. Any unresolved toxicities from prior therapy greater than National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAEv5.0) Grade 1, at the time of screening except for alopecia
6. Inability to swallow the study medication, any seriously (NCI-CTCAEv5.0 ≥ Grade 3) chronic gastrointestinal disorder, malabsorption syndrome or any other conditions with influence on gastrointestinal absorption
7. Active central nervous system metastases
8. Any active infection which has not been controlled at screening

Other exclusion criteria apply for participating in the Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Pre-dose up to approximately 32 months post-dose

SECONDARY OUTCOMES:
Duration of Response (DoR) | Pre-dose up to approximately 32 months post-dose
Disease Control Rate (DCR) | Pre-dose up to approximately 32 months post-dose
Progression Free Survival (PFS) | Pre-dose up to approximately 32 months post-dose
Time to Tumor Progression (TTP) | Pre-dose up to approximately 32 months post-dose
Time to Response (TTR) | Pre-dose up to approximately 32 months post-dose
Time to Treatment Failure (TTF) | Pre-dose up to approximately 32 months post-dose
Overall Survival (OS) | Pre-dose up to approximately 32 months post-dose
1-year Progression Free Survival | Pre-dose up to 1 year post-dose
  Ratio of participants who do not have objective tumor progression or have not died 1 year after the first dose of IP.
1-year Survival | Pre-dose up to 1 year post-dose
  Ratio of surviving participants 1 year after the first dose of IP.
Area Under The Curve (AUC) of Sutetinib Maleate Capsule | Pre-dose up to 24 hours post-dose
Maximum Plasma Concentration (Cmax) of Sutetinib Maleate Capsule | Pre-dose up to 24 hours post-dose
Minimum Plasma Concentration (Cmin) of Sutetinib Maleate Capsule | Pre-dose up to 24 hours post-dose
Time to Peak Drug Concentration (Tmax) of Sutetinib Maleate Capsule | Pre-dose up to 24 hours post-dose
Sutetinib Maleate Capsule half-life (T1/2) | Pre-dose up to 24 hours post-dose
Apparent Clearance (CL/f) of Sutetinib Maleate Capsule | Pre-dose up to 24 hours post-dose
Volume of Distribution (Vz/F) of Sutetinib Maleate Capsule | Pre-dose up to 24 hours post-dose
Number of Participants Experiencing Adverse Events (AE) | Pre-dose up to approximately 32 months post-dose
Number of Participants Experiencing Adverse Drug Reactions (ADR) | Pre-dose up to approximately 32 months post-dose
Number of Participants Experiencing Serious Adverse Events (SAE) | Pre-dose up to approximately 32 months post-dose
Number of Participants Experiencing Srious Adverse Reactions (SAR) | Pre-dose up to approximately 32 months post-dose

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Oncology Physicians Network Healthcare, Glendale, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Moffitt Cancer Center, Tampa, Florida
  - University Cancer & Blood Center (UCBC) - Athens, Athens, Georgia
  - Mission Cancer + Blood - Mission Cancer Foundation, Des Moines, Iowa
  - Norton Cancer Institute - Downtown, Louisville, Kentucky
  - Northwell Health, New Hyde Park, New York
  - Perlmutter Cancer Center - 34th Street, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No